CLINICAL TRIAL: NCT01588860
Title: Mutation Analysis and Copy Number Changes of KRAS and BRAF Gene in Taiwanese Cases of Biliary Tact Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 099084-F
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2010-12

CONDITIONS: Biliary Tract Adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Fixed tissue in the paraffin embedded blocks
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Cholangiocarcinoma is a fatal malignant neoplasm originating from biliary tracts and constitutes about 5-10% of primary liver cancers, characterized by a poor prognosis. High prevalence in southeast and eastern Asia has been observed. At present, the cellular and molecular mechanisms leading to oncogenesis of cholangiocarcinoma remain unclear.

The RAS gene product has a key role in controlling cell growth and differentiation through its intrinsic GTPase activity. Point mutations that activate the RAS protein and its downstream cascade have been observed in human tumors. Both KRAS and BRAF are members of the RAS-RAF-MEK-ERK-MAP kinase pathway which mediates cellular response to growth signals. Somatic KRAS mutations are found at high rates in leukemia, colon cancer, pancreatic cancer and lung cancer. Studies from European and Japanese groups have recently described that activating KRAS/ BRAF mutations may play a role in the carcinogenesis of cholangiocarcinoma of the biliary tracts, but our preliminary data demonstrated low frequency of KRAS and BRAF mutation in the same tumor as well as the results from Thailand. In this study, the investigators hypothesize copy number changes rather than genetic mutation of either KRAS or BRAF genes may be the key findings of Taiwanese cases of the adenocarcinoma from the biliary tracts.

ELIGIBILITY:
Inclusion Criteria:

* The patients diagnosed as biliary tact adenocarcinoma.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients diagnosed as biliary tact adenocarcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pathology, Far Eastern Memorial Hospital and National Taiwan University Hospital, Taipei, Taiwan